CLINICAL TRIAL: NCT06878313
Title: Role of Elastic Power in Acute Respiratory Distress Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Nestor Pistillo, Head of intensive care, Hospital El Cruce
Other Study IDs: UTIA El Cruce
Record Dates: First submitted 2025-03-11; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: ARDS (Moderate or Severe); Adult Patients
Keywords: ARDS; VILI; Mechanical Ventilation
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Mechanical ventilation is essential for managing acute respiratory distress syndrome (ARDS), but it can also cause ventilator-induced lung injury (VILI) due to mechanical forces. VILI results from the interaction between lung structure and mechanical ventilation factors, such as tidal volume, plateau pressure, driving pressure, inspiratory flow, respiratory rate, and PEEP. Intrinsic factors like lung heterogeneity further increase the risk.

Elastic power (EP), a key component, is linked to repetitive alveolar stretching and disease progression.

Study Objectives:

Examine the correlation between elastic power and pulmonary hyperinflation. Compare EP's sensitivity and specificity with other overdistension markers like driving pressure, plateau pressure, upper inflection point, and compliance.

DETAILED DESCRIPTION:
Introduction:

Mechanical ventilation is a fundamental intervention in the management of acute respiratory distress syndrome (ARDS), providing life support while the lungs recover. However, it can also induce ventilator-induced lung injury (VILI) due to the mechanical forces applied during ventilation.

VILI arises from the interaction between lung structure-mainly composed of elastin and collagen fibers embedded in a hydrated extracellular matrix-and the mechanical factors imposed by ventilation. Among these, tidal volume (Vt), plateau pressure (PPlat), driving pressure (∆P), inspiratory flow (Ṹ), respiratory rate (RR), and, in certain cases, positive end-expiratory pressure (PEEP) have been identified as key determinants of lung injury. Additionally, intrinsic factors such as lung heterogeneity and reduced ventilatory capacity may increase the risk of VILI even under protective ventilation strategies.

The positive pressure generated by mechanical ventilation is distributed between the lungs and the thoracic cage. The pressure applied directly to the lungs is known as transpulmonary pressure (Ptp), defined as the difference between alveolar pressure and pleural or esophageal pressure. Ptp expands the alveoli until it balances the tension of the alveolar wall, which opposes this expansion. Alveolar wall tension directly depends on the surface tension of the liquid lining the alveoli. Under normal conditions, pulmonary surfactant reduces alveolar surface tension. However, in ARDS, inflammation and alveolar damage degrade and inhibit surfactant production, increasing surface tension, promoting alveolar collapse and stiffness.

Although the terms "pressure" and "tension" may seem synonymous, the relationship between intra-alveolar pressure and alveolar wall tension is non-linear, as described by Laplace's law:

Tension= Pressure × Radius / 2 × Thickness

This implies that, under the same Ptp, ventral alveoli (larger and with thinner walls) experience greater deformation and tension than dorsal alveoli (smaller and with thicker walls). In this context, if alveolar deformation exceeds the structural tolerance threshold, it can lead to microfractures, pulmonary edema, hemorrhage, and inflammatory activation, contributing to multiple organ dysfunction and increased mortality.

Although alveolar tension cannot be directly measured in clinical settings, tools such as computed and electrical impedance tomography allow for indirect estimation of alveolar overdistension risk. Without airflow, alveolar tension varies between a baseline value-determined by PEEP-and a maximum value at end-inspiration-defined by PPlat. Thus, lung stress can be expressed as:

Stress (ΔPtp)= Ptp at end-inspiration-Ptp at end-expiration\text

However, lung stress and strain are static variables that do not fully capture the dynamic changes occurring during the ventilatory cycle. Animal studies have shown that VILI correlates with flow magnitude, suggesting that higher deformation rates reduce the alveolus's ability to adapt. This phenomenon is described by the Kelvin-Voigt equation for viscoelastic materials:

Stress= k × Strain + η × Strain Rate

where k represents the Young's modulus of elasticity and η the viscosity modulus.

Since VILI results from a combination of pressure, volume, and flow, mechanical power emerges as an integrative concept that expresses these variables in terms of energy per unit of time. It is estimated that a mechanical power exceeding 12 J/min surpasses the lung's adaptive capacity, increasing the risk of VILI and mortality in ARDS. Among its components, elastic power (EP) is responsible for repetitive alveolar stretching and appears to be most directly associated with ARDS severity.

Study Objectives:

1. To evaluate whether elastic power correlates with pulmonary hyperinflation.
2. To compare the sensitivity and specificity of elastic power with other overdistension markers, such as driving pressure (∆P), plateau pressure (PPlat), the upper inflection point of the V/P curve, and respiratory system compliance (CRS).

Materials and Methods:

Ethical Considerations: The study requires evaluation and subsequent approval from the institution's ethics and research committee, following the principles established in the Declaration of Helsinki. The study was registered on ClinicalTrials.gov before patient inclusion. Inclusion in the study requires prior informed consent authorization from an adult family member.

Inclusion Criteria: Adult patients (≥18 years) with moderate to severe ARDS, according to the Berlin expert consensus definition, will be prospectively and consecutively included.

Exclusion Criteria: Patients will be excluded if they meet any of the following criteria:

History of emphysema, asthma, or pneumothorax. Severe instability at the time of the study that would prevent the recruitment maneuver, defined by at least one of the following indicators: SaO2 ≤ 90%, shock requiring more than 0.5 γ/kg/min of norepinephrine, complex arrhythmia, myocardial ischemia, or intracranial hypertension unresponsive to first-line measures.

Patients with do-not-resuscitate orders or pregnant women. Procedure: Under deep sedation and analgesia (Cambridge-Ramsay: V to VI) and using neuromuscular blocking agents, patients will be ventilated in the supine position using a ventilator (SERVO-s, Maquet, Germany) in volume control mode (VCV) with a tidal volume of 6 ml/kg of predicted body weight (PBW), a respiratory rate of 18 breaths per minute, and a constant flow.

After performing a gentle aspiration of airway secretions using a closed circuit, PEEP titration will begin stepwise, increasing in increments of 2 cmH2O starting from 8 cmH2O (baseline condition), progressively increasing until a maximum of 20 cmH2O or a plateau pressure of 45 cmH2O is reached, whichever occurs first.

At each PEEP level, respiratory mechanics, vital parameters, and impedance tomography images will be evaluated after a short stabilization period of the studied variables.

Finally, after determining the optimal PEEP based on the best respiratory system compliance (CRS), PEEP will be titrated 2 cmH2O above its optimal value to prevent alveolar derecruitment and improve patient safety.

Criteria for Stopping the Procedure: These include SaO2 below 85%, complex arrhythmias, or hemodynamic instability (mean arterial pressure <60 mmHg).

Measurement of Transpulmonary Pressures: Since direct measurement of pleural pressure (Ppl) is complicated in clinical practice, esophageal pressure (Pes) was used as a surrogate. An inflatable balloon catheter will be inserted into the lower third of the esophagus while the patient remains in the supine position, according to standard technique. The balloon will be inflated with the minimum volume of air necessary to ensure accurate pressure recordings.

Transpulmonary pressure (Ptp) measurements will be obtained using a respiratory mechanics monitoring system (FluxMed GrT, Buenos Aires, Argentina).

Electrical Impedance Tomography (EIT): EIT is a medical imaging technology that detects impedance changes through specific image algorithms by applying low-intensity electrical currents and measuring surface voltages via electrodes placed around the chest.

In this study, continuous signal recording will be performed using the commercial device with 32 electrodes, Infivision ET1000 (Infivision Medical Imaging Technology Co., Ltd., Beijing, China). This device allows non-invasive assessment of both ventilation and perfusion in four lung regions of interest (ROIs), defined by horizontal lines within the thoracic contour: ROI 1 (ventral), ROI 2 (central ventral), ROI 3 (central dorsal), and ROI 4 (dorsal).

Perfusion signals will be extracted using frequency domain filtering techniques. By analyzing the signal spectrum, the cardiac signal (which occurs at higher frequencies than the respiratory signal) will be isolated using a digital bandpass filter. Areas identified as hyperinflated will be quantified as a percentage relative to the respective ROI.

Evaluation of Elastic Power:

Elastic Power (EP): EP = 0.098 × RR × [(Vt × PEEP) + (Vt × ΔP) / 2].

ELIGIBILITY:
Inclusion Criteria: Adult patients (≥18 years) with moderate-to-severe acute respiratory distress syndrome (ARDS), as defined by the Berlin criteria, were prospectively and consecutively included.

-

Exclusion Criteria: Patients were excluded if they met at least one of the following criteria:

* History of emphysema, asthma, or pneumothorax.
* Severe instability at the time of the study preventing the PEEP titration maneuver, defined by at least one of the following indicators: SaO₂ ≤ 90%, shock requiring >0.5 γ/kg/min of norepinephrine, complex arrhythmia, myocardial ischemia, or intracranial hypertension refractory to initial treatment.
* Patients with do-not-resuscitate orders and pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with moderate-to-severe acute respiratory distress syndrome (ARDS) included in UCI.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between pulmonary hyperinflation and pulmonary elastic power | 1 hour

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie Y, Shi J, Liu S, Chen X, Wang Y, Li X, Yan Y. Association of elastic power in mechanical ventilation with the severity of acute respiratory distress syndrome: a retrospective study. Eur J Med Res. 2024 Jan 3;29(1):5. doi: 10.1186/s40001-023-01577-7. PMID 38173033
- [Background] Modesto I Alapont V, Aguar Carrascosa M, Medina Villanueva A. Stress, strain and mechanical power: Is material science the answer to prevent ventilator induced lung injury? Med Intensiva (Engl Ed). 2019 Apr;43(3):165-175. doi: 10.1016/j.medin.2018.06.008. Epub 2018 Nov 5. No abstract available. English, Spanish. PMID 30409677
- [Background] Marini JJ, Thornton LT, Rocco PRM, Crooke PS. From pressure to tension: a model of damaging inflation stress. Crit Care. 2023 Nov 15;27(1):441. doi: 10.1186/s13054-023-04675-4. PMID 37968744
- [Background] Gattinoni L, Marini JJ, Collino F, Maiolo G, Rapetti F, Tonetti T, Vasques F, Quintel M. The future of mechanical ventilation: lessons from the present and the past. Crit Care. 2017 Jul 12;21(1):183. doi: 10.1186/s13054-017-1750-x. PMID 28701178